CLINICAL TRIAL: NCT02187406
Title: Ankle Athletic Taping Fatigue After a Standard Tennis Warm up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CEU-007
Record Dates: First submitted 2014-07-03; First posted 2014-07-11 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Ankle Injuries
Keywords: athletic tape; tennis; warm-up exercise
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Traditional ankle athletic taping (Experimental): Described by Purcell and Schuckman (2009)
  Interventions: Procedure: Traditional ankle athletic taping
- modified ankle athletic taping (Experimental): Described by Montag and Asmussen (1992)
  Interventions: Procedure: Modified ankle athletic taping

INTERVENTIONS:
Procedure: Modified ankle athletic taping
  Arms: modified ankle athletic taping
Procedure: Traditional ankle athletic taping
  Arms: Traditional ankle athletic taping

SUMMARY:
Identify, quantify and compare the fatigue caused in two ankle athletic tapes after the completion of a tennis warm-up.

ELIGIBILITY:
Inclusion Criteria:

* There have been no ankle injury in the last 6 months (defined as any problem ankle injury that limited normal activity for more than 48 hours).
* Not having any neurological, circulatory or degenerative disease or to upset the balance in the lower limbs.
* Not having had any fractures or have undergone surgery on the lower limbs.
* No experience pain in the ankle at the time of the study.

Exclusion Criteria:

* Allergy to any of the materials used bandage
* Suffer an injury before taking the last measurement that prevented them from developing their sport normally.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in the Goniometry of the active range of movement | participants will be followed for the duration of a standard tennis Warm up, an expected average of 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Francisco García-Muro San José, MSc, PT, Study Director — San Pablo CEU University; Serafín Álvarez Álvarez, MSc, PT, Principal Investigator — San Pablo CEU University; Luis Fernández Rosa, Phd, MD, Study Chair — San Pablo CEU University
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain